CLINICAL TRIAL: NCT05300568
Title: Women's Treatment Preferences for Moderate to Severe Vasomotor Symptoms (VMS) (WARMER Study)
Brief Title: A Survey About Trade-offs When Choosing Menopause Treatments
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2693-MA-3237
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Moderate to Severe Vasomotor Symptoms
Keywords: menopause; vasomotor symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- post-menopausal women: post-menopausal women with moderate to severe VMS associated with menopause
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-product related survey.

SUMMARY:
This study is an online survey of women in menopause with moderate to severe hot flashes. Menopause, a normal part of life, is the time after a woman's last period. Hot flashes often occur during menopause. They can disrupt a woman's daily life.

This study is about collecting information only. There will be no treatment in this study. This study will provide information on the trade-offs women are willing to make when deciding which treatment or treatments work best for them.

Women from Australia, Canada, Denmark, France, Germany, Italy, Spain, Sweden and the United Kingdom (UK) will take part in this study.

Women will be recruited through a third-party recruitment company.

Most women will be asked to complete an online survey. Before the survey is sent to the women in the study, it will be tested by a small group of women. This group will be asked to take part in a telephone interview while taking the survey. They will be asked to say their thoughts aloud while completing the survey. Researchers will record this and also take notes. The aim of the interview is to check that the survey is understood by the women before it is sent out to the rest of the women.

The survey will have 3 sections: Firstly, the women will answer questions about their experience with menopause and their symptoms. Next, they will be shown pros and cons for specific treatments for their menopause symptoms. The women will be asked to choose which treatment they would prefer, based on this information. Finally, they will answer questions on how their menopause symptoms have impacted their lives.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Australia, Canada, Denmark, France, Germany, Italy, Spain, Sweden, or the United Kingdom
* Experience at least 14 moderate or severe VMS episodes associated with menopause per week (or 2 to 3 episodes per day)
* Self-reported completion of natural menopause (post-menopausal)
* Willing and able to provide consent to take part in the study; Speak native language of country of participation
* Telephone interview only: Willing and able to participate in a telephone interview, and be audio recorded

Exclusion Criteria:

* Experienced treatment related menopause either as a result of medical or surgical intervention
* Difficulty understanding or communicating in the language(s) of Australia, Canada, Denmark, France, Italy, Spain, Sweden, or the United Kingdom
* Online survey only: Participation in the Telephone interview

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-menopausal women with moderate to severe VMS associated with menopause
Sampling Method: Non-Probability Sample
Enrollment: 1465 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-27 (Actual)

PRIMARY OUTCOMES:
Part-worth utilities for each treatment attribute | 1 day (once through survey)
  The effect of changes in each attribute on preferences.
  Participants' preferences for Vasomotor Symptoms (VMS) treatment attributes will be collected via a discrete choice experiment (DCE).
  Participants will be asked to choose their preferred option among two treatments or no treatment.
  Negative part-worth utility indicates less desired levels and positive part-worth utility indicates more desired levels of attributes.
Relative attribute importance scores | 1 day (once through survey)
  Relative attribute importance scores will be derived from part-worth estimates and measure the maximum percentage contribution to a preference that relates to a change in each attribute.
Maximum acceptable risk | 1 day (once through survey)
  Maximum acceptable risk will be derived from part-worth estimates and measures how much risk (i.e., for each included risk) participants are willing to accept for a one-unit change in each other attribute.
Minimum acceptable benefit | 1 day (once through survey)
  Minimum acceptable benefit will be derived from part-worth estimates and measures the minimum acceptable reduction in the frequency of VMS for a unit change in each other attribute.

SECONDARY OUTCOMES:
Estimated probability that a specific treatment profile will be chosen | 1 day (once through survey)
  A set of treatment profiles will be generated using the attributes included in the discrete choice experiment (DCE). The probability of each profile being selected will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Study Director — Astellas Pharma Europe Ltd.
Locations (1):
- Site GB44001, Hammersmith, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.